CLINICAL TRIAL: NCT04839289
Title: A Study to Compare Patient Perceptions of Two Different Hearing Aid Signal Processing Philosophies
Brief Title: Hearing Aid Signal Processing Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-311
Record Dates: First submitted 2021-02-25; First posted 2021-04-09 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Masking Description: Identifying information will be removed from the hearing instruments before fitting the participants. However, participants may be able to research hearing instruments and identify devices based on physical appearance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- A-B-A (Experimental): Participants will be fit with hearing instruments A and B in the following order:
  Hearing instrument A Hearing instrument B Hearing instrument A
  Interventions: Device: Receiver-in-canal hearing instrument; Manufacturer A; Device: Receiver-in-canal hearing instrument; Manufacturer B
- B-A-B (Experimental): Participants will be fit with hearing instruments A and B in the following order:
  Hearing instrument B Hearing instrument A Hearing instrument B
  Interventions: Device: Receiver-in-canal hearing instrument; Manufacturer A; Device: Receiver-in-canal hearing instrument; Manufacturer B

INTERVENTIONS:
Device: Receiver-in-canal hearing instrument; Manufacturer A — Commercially available receiver-in-canal hearing instrument from manufacturer A
Device: Receiver-in-canal hearing instrument; Manufacturer B — Commercially available receiver-in-canal hearing instrument from manufacturer B

SUMMARY:
Participants will be fit with each of two hearing instruments in an ABA cross-over design. The study will consist of a total of three approximately 10-day home trials with the devices. Participants will be asked to provide qualitative feedback to investigators regarding the performance of and their preference for each hearing instrument.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe sensorineural hearing loss
* Current hearing aid user

Exclusion Criteria:

* Lack of willingness to wear study devices for approximately one month
* Inability to travel to study appointments or to complete questionnaires.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- A-B-A: Participants will be fit with hearing instruments A and B in the following order:
  Hearing instrument A Hearing instrument B Hearing instrument A
  Receiver-in-canal hearing instrument; Manufacturer A: Commercially available receiver-in-canal hearing instrument from manufacturer A
  Receiver-in-canal hearing instrument; Manufacturer B: Commercially available receiver-in-canal hearing instrument from manufacturer B
- B-A-B: Participants will be fit with hearing instruments A and B in the following order:
  Hearing instrument B Hearing instrument A Hearing instrument B
  Receiver-in-canal hearing instrument; Manufacturer A: Commercially available receiver-in-canal hearing instrument from manufacturer A
  Receiver-in-canal hearing instrument; Manufacturer B: Commercially available receiver-in-canal hearing instrument from manufacturer B
Period: Overall Study
Arm/Group | A-B-A | B-A-B
Started | 18 | 9
Completed | 17 | 9
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-B-A | B-A-B | Total
Number analyzed (Participants) | 17 | 9 | 26
Age, Continuous [Mean (Full Range); unit: years] | 73.5 [59 to 88] | 67 [60 to 77] | 70.25 [59 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 9 | 3 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 0 | 17
  China | 0 | 9 | 9
Mild to moderate severe sensorineural hearing loss, bilaterally [Number; unit: participants] | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Standardized Validated Questionnaire Measuring Hearing Aid Sound Quality for First Study Set Worn, i.e. Study Set A for Arm A-B-A and Study Set B for Arm B-A-B
Description: Qualitative feedback questionnaire to gather feedback on particular areas of focus. Subjects will rate hearing performance and sound quality on a Likert scale with lowest number equivalent to worst performance or worst sound quality (1) and higher number equivalent to best performance or best sound quality (10).
Time Frame: End of home trial 1 (Day 10 of study)
Population: Participants who were fit with first set of hearing aids for first home trial. For arm A-B-A, the outcomes will measure hearing aid A, and for arm B-A-B, the outcomes will measure hearing aid B
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-B-A | B-A-B
Number analyzed (Participants) | 17 | 9
score on a scale | 7.16 (0.46) | 7.12 (0.85)

2. Primary Outcome: Standardized Validated Questionnaire Measuring Hearing Aid Sound Quality for Second Study Set Worn, i.e. Study Set B for Arm A-B-A and Study Set A for Arm B-A-B
Description: as for outcome 1
Time Frame: End of home trial 2 (20 days after study start)
Population: Participants who were fit with second set of hearing aids for second home trial. For arm A-B-A, the outcomes will measure hearing aid B, and for arm B-A-B, the outcomes will measure hearing aid A
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-B-A | B-A-B
Number analyzed (Participants) | 17 | 9
score on a scale | 7.61 (0.42) | 6.70 (0.98)

3. Primary Outcome: Standardized Validated Questionnaire Measuring Hearing Aid Sound Quality for Third Study Set Worn, i.e. Study Set A for Arm A-B-A and Study Set B for Arm B-A-B
Description: as for outcome 1
Time Frame: End of home trial 3 (30 days after study start)
Population: Participants who were fit with third set of hearing aids for third home trial. For arm A-B-A, the outcomes will measure hearing aid A, and for arm B-A-B, the outcomes will measure hearing aid B
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-B-A | B-A-B
Number analyzed (Participants) | 17 | 9
score on a scale | 7.28 (.51) | 7.52 (0.95)
Statistical Analysis 1: Comparison: A-B-A; Null hypothesis: Subjective ratings of sound quality would not be different between any of the three study hearing aids when measured with a validated sound quality questionnaire. Analysis was done after all three home trials completed so all three sets of study devices could be compared; Test type: Other; p > 0.05, t-test, 2 sided — When p-value is adjusted for multiple comparisons, the level of statistical significance must be </= to .01666667 (.05/3)
Statistical Analysis 2: Comparison: B-A-B; [analysis description as in outcome 3, analysis 1]; Test type: Other; p < .0167, t-test, 2 sided — [p-value comment as in outcome 3, analysis 1]

4. Primary Outcome: Standard Validated Questionnaire Measuring Satisfaction of Hearing Aid Performance and Features for First Study Set Worn.
Description: Measures satisfaction on various aspects of hearing aid use on a scale from 1 to 5, with 1 = Very unsatisfied to 5 = Very satisfied, and 3 = Neutral.
  .
Time Frame: End of home trial 1 (Day 10 of study)
Population: Participants who were fit with first set of hearing aids for first home trial. For arm A-B-A, the outcomes will measure study set A, and for arm B-A-B, the outcomes will measure study set B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-B-A | B-A-B
Number analyzed (Participants) | 17 | 9
score on a scale | 3.94 (0.59) | 3.80 (.30)

5. Primary Outcome: Standard Validated Questionnaire Measuring Satisfaction of Hearing Aid Performance and Features for Second Study Set Worn.
Description: Measures satisfaction on various aspects of hearing aid use on a scale from 1 to 5, with 1 = Very unsatisfied to 5 = Very satisfied, and 3 = Neutral.
Time Frame: End of home trial 2 (Day 20 of study)
Population: Participants who were fit with second set of hearing aids for second home trial. For arm A-B-A, the outcomes will measure study set B, and for arm B-A-B, the outcomes will measure study set A.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-B-A | B-A-B
Number analyzed (Participants) | 17 | 9
score on a scale | 4.24 (0.54) | 3.76 (0.28)

6. Primary Outcome: Standard Validated Questionnaire Measuring Satisfaction of Hearing Aid Performance and Features for Third Study Set Worn.
Description: as for outcome 5
Time Frame: End of home trial 3 (Day 30 of study)
Population: Participants who were fit with third set of hearing aids for third home trial. For arm A-B-A, the outcomes will measure study set A, and for arm B-A-B, the outcomes will measure study set B.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-B-A | B-A-B
Number analyzed (Participants) | 17 | 9
score on a scale | 4.12 (0.47) | 3.99 (0.21)
Statistical Analysis 1: Comparison: A-B-A; Null hypothesis: Satisfaction with hearing aid performance and features would not be different between any of the three study hearing aids when measured with subjective hearing aid satisfaction questionnaire. Analysis was done after all three home trials completed so all three sets of study devices could be compared; Test type: Other; p < .01666667, t-test, 2 sided — When p-value is adjusted for multiple comparisons, the value must be </= to .01666667 (.05/3)
Statistical Analysis 2: Comparison: B-A-B; [analysis description as in outcome 6, analysis 1]; Test type: Other; p < .01666667, t-test, 2 sided — When adjusted for multiple comparisons, the p-value must be </= to .01666667 (.05/3)

ADVERSE EVENTS:
Time Frame: The time frame in which the participant was enrolled in the study which was up to 8 weeks.
Groups:
- Receiver-in-canal Hearing Instrument Manufacturer A: All participants who received Manufacturer A study set A during the course of the trial
  Receiver-in-canal hearing instrument; Manufacturer A: Commercially available receiver-in-canal hearing instrument from manufacturer A
  Receiver-in-canal hearing instrument; Manufacturer B: Commercially available receiver-in-canal hearing instrument from manufacturer B
- Receiver-in-canal Hearing Instrument Manufacturer B: All participants who received Manufacturer B study set B during the course of the trial
  Receiver-in-canal hearing instrument; Manufacturer A: Commercially available receiver-in-canal hearing instrument from manufacturer A
  Receiver-in-canal hearing instrument; Manufacturer B: Commercially available receiver-in-canal hearing instrument from manufacturer B
Arm/Group | Receiver-in-canal Hearing Instrument Manufacturer A | Receiver-in-canal Hearing Instrument Manufacturer B
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT04839289/Prot_SAP_000.pdf